CLINICAL TRIAL: NCT06139653
Title: Therapeutic Effects of CardioBreath Aplication Versus Inspiratory Muscle Training (IMT) on Vagal Cardiac Modulation, Pulse Wave Velocity Maximal Respiratory Pressures in Heart Failure Patients: Cross-over Randomized Control Trial
Brief Title: CardioBreathApp vs IMT in Heart Failure
Acronym: CardioBreath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UP6065/23
Record Dates: First submitted 2023-08-31; First posted 2023-11-18 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-12

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Sequential Assignment The participants will be randomized into 2 intervention groups as follows: Group 1: Moment 1: IMT Moment 2: CardioBreath®App. Group 2: Moment 1: CardioBreath®App Moment 2: IMT. The intervention will long five weeks. The exercises will be performed at home for five days/week
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) Participants will not know about other arms. Outcome assessors will not know the arms participant belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - IMT CB (Active Comparator): Moment 1: IMT and moment 2: CardioBreath. Participants will have PowerBreath device for IMT adjusted for 30% with weekly adjustment of maximal inspiratory pressure and will perform the exercise at home for five days/week. They will perform 5 sets of 10 repetitions twice a day for five weeks.
  CardioBreathApp group will have the app settings of profile and spontaneous respiratory rate to determine the exercise rate of exercises, which will be performed at home for five days/week during 5 sets of one minute with 30' of rest between the sets twice a day. respiratory rate of exercise will be determined by 80% of spontaneous respiratory rate twice a day for five weeks. An once a week meeting will provide readjustment of respiratory rate to perform exercises. One week washout will be taken between the two interventions in order to cleanse motor memory of respiratory act.
  Interventions: Device: Moment 1: IMT. Moment 2 CardioBreath.
- Group 2 - CB IMT (Active Comparator): Moment 1: CardioBreath and moment 2: IMT. Participants will have PowerBreath device for IMT adjusted for 30% with weekly adjustment of maximal inspiratory pressure and will perform the exercise at home for five days/week. They will perform 5 sets of 10 repetitions twice a day for five weeks.
  CardioBreathApp group will have the app settings of profile and spontaneous respiratory rate to determine the exercise rate of exercises, which will be performed at home for five days/week during 5 sets of one minute with 30' of rest between the sets twice a day. respiratory rate of exercise will be determined by 80% of spontaneous respiratory rate twice a day for five weeks. An once a week meeting will provide readjustment of respiratory rate to perform exercises. One week washout will be taken between the two interventions in order to cleanse motor memory of respiratory act.
  Interventions: Device: Moment 1: CardioBreath and moment 2: IMT.

INTERVENTIONS:
Device: Moment 1: IMT. Moment 2 CardioBreath. — Participants will have PowerBreath device for IMT adjusted for 30% with weekly adjustment of maximal inspiratory pressure and will perform the exercise at home for five days/week. They will perform 5 sets of 10 repetitions twice a day for five weeks.
  CardioBreathApp group will have the app settings of profile and spontaneous respiratory rate to determine the exercise rate of exercises, which will be performed at home for five days/week during 5 sets of one minute with 30' of rest between the sets twice a day. respiratory rate of exercise will be determined by 80% of spontaneous respiratory rate twice a day for five weeks. An once a week meeting will provide readjustment of respiratory rate to perform exercises. One week washout will be taken between the two interventions in order to cleanse motor memory of respiratory act.
  Arms: Group 1 - IMT CB
Device: Moment 1: CardioBreath and moment 2: IMT. — CardioBreathApp group will have the app settings of profile and spontaneous respiratory rate to determine the exercise rate of exercises, which will be performed at home for five days/week during 5 sets of one minute with 30' of rest between the sets twice a day. respiratory rate of exercise will be determined by 80% of spontaneous respiratory rate twice a day for five weeks. An once a week meeting will provide readjustment of respiratory rate to perform exercises. One week washout will be taken between the two interventions in order to cleanse motor memory of respiratory act.
  Participants will have PowerBreath device for IMT adjusted for 30% with weekly adjustment of maximal inspiratory pressure and will perform the exercise at home for five days/week. They will perform 5 sets of 10 repetitions twice a day for five weeks.
  Arms: Group 2 - CB IMT

SUMMARY:
Heart failure (HF) is a systemic clinical syndrome defined as cardiac dysfunction, which causes inadequate blood supply to meet metabolic needs. One of the most expressive markers of HF is neurologic exacerbation, with expected sympathetic hyperactivation, increased activity of the renin-angiotensin-aldosterone system and elevation of vasopressin levels. These changes compensate the low cardiac output in the onset of ventricular dysfunction ensure a long term high blood perfusion pressure,though aggravate this dysfunction and contributes to the HF progression. There are evidences ofthe therapeutic effects of respiratory exercise techniques for HF patients. However, it demands new data for larger prescription and employment of these kind of exercises. Advanced technologies allowed the elaboration of the application for slow breathing CardioBreath. So far, it requires the possibility of comparison of their effects versus widely validated Inspiratory Muscle Trainig (IMT) on respiratory and cardiovascular outcomes in order to elucidate their specific benefits. In this way compare CardioBreath ® App versus IMT through a crossover randomized clinical trial design may elucidate the response effects of these interventions in these patients.

DETAILED DESCRIPTION:
The impact of pulmonary, ventilatory and cardiovascular impairment in patients with congestive heart failure (CHF) highlights the therapeutic relevance of breathing exercises for these functions. In addition, other benefits such as lowering blood pressure,increased cardiac vagal modulation, improved vascular function and psychosocial handling (anxiety, depression and stress) may be expected. Inspiratory Muscle Training (IMT) and slow yoga breathing are widely endorsed as beneficial by a large amount of evidence. The newly developed app CardioBreath ® is based on a breathing technique of yoga (ujjayi pranayama) through respiratory rates (RR) slower than the user's spontaneous RR, in a set of strategies with pedagogical prescription, guidance and monitoring of this type of exercises. This study aims to compare IMT exercises with those of the CardioBreath ® application on , strength respiratory muscle (manuvacuometry), cardiac vagal modulation (heart rate variability), arterial stiffness (heart rate wave velocity) and diaphragm thickness in CHF patients after their hospital discharge in Institute of Cardiology of Rio Grande do Sul. Methods: Crossover randomized control trial will recruit post-discharge CHF patients who will be evaluated through, Finometer system (HR and BP variability/cardiac vagal modulation), Arterial Stiffness (oscillometric method), for indexes of central arterial pressure, velocity pulse waveform (large artery stiffness) and Aix 75 (small artery stiffness), Respiratory Muscle Strength by Manovacuometry and Diaphragm Thickness by ultrasound. Patients will be randomized to two orders of intervention Group 1- Moment 1 TMI and Moment 2 CardioBreath App Group 2- Moment 1 CardioBreath App and Moment 2 TMI. The interventions will face-to-face assistance once a week for intensity adjustments, with 5 sets of 10 repetitions twice a day during week days for five weeks both for CardioBreath and IMT. Patients will be evaluated immediately after hospital discharge and at the end of the Moment 1, they will carry out a washout period of one week between the moments 1 and 2 and new evaluations before and after moment 2. The data obtained will be analyzed by intention to treat (ITT) and presented as means (M) ± standard deviation (SD). Will be tested for normality through the test by Shapiro Wilk. Differences between interventions will be detected through Student's t-test for paired samples. Correlations between variables will be obtained by Pearson's correlations for parametric and Spearman for non-parametric data, with significance level p< 0.05. Expected Results: Although there is no data comparing IMT and slow breathing in CHF patients, significant results are expected in the two intervention groups, and differences between both protocols will point to their specific applicability.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive CHF patients in treatment at the outpatient clinic (Institute of Cardiology)
* Of both sexes
* Aged between 40 and 70 years
* And ejection fraction (EF) reduced (<40%)
* Who have access to a mobile device with access to Internet.

Exclusion Criteria:

* active smoking
* BMI <30
* Diagnosis of sleep apnea
* Heart failure of congenital origin
* Valve disease.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular autonomic control by heart rate variability(HRV) | Time Frame: 30 minutes
  High Frequency (HF) component of HRV (ms2 = squared milliseconds) as measure of vagal modulation acquired by Finometer and analyzed by Cardioseries Software.
High Frequency (HF) component of HRV (ms2 = squared milliseconds) as measure of vagal modulation. | 30 minutes
  Heart rate variability collected by Polar V800 device and analyzed by Kubios Software. The 10 minutes assessment (concomitant with the Finometer acquisition) either for 5 weeks interventions and also in acute mode of 5 minutes of slow breathing of 10 cycles per minute (baseline 10 minutes/ 5 minutes slow breathing/ 10 minutes post intervention).

SECONDARY OUTCOMES:
Respiratory rate by Pneumotrace respiratory belt | 30 minutes along with Finometer
  Respiratory rate in cycles per minute (CPM)

OTHER OUTCOMES:
Carotid -femoral pulse wave velocity (VOP) | 15 minutes
  Arterial Stiffness (oscillometric method - Arteris)
Diaphragm Thickness by ultrasound | 5 minutes
  Increase diaphragm thickness (mm)
Strength Respiratory Muscle | 10 minutes
  Manuvacuometry

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Institute of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No